CLINICAL TRIAL: NCT04311281
Title: [F-18] FDDNP-PET Clinical Protocol for Visualizing Brain Proteinopathies to Assist in the Diagnosis of Persons With Suspected Chronic Traumatic Encephalopathy and Alzheimer's Disease
Brief Title: FDDNP Protocol for Visualizing Brain Proteinopathies to Assist in the Diagnosis of Persons With Suspected CTE and AD
Acronym: FDDNP
Status: Withdrawn | Type: Observational
Why Stopped: Insufficient Funding
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Helen Lavretsky, MD, Principal Investigator, University of California, Los Angeles
Other Study IDs: 18-001176
Record Dates: First submitted 2020-03-12; First posted 2020-03-17 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Suspected Chronic Traumatic Encephalopathy (CTE) or Traumatic Encephalopathy Syndrome (TES); Suspected Alzheimer's Disease (AD)
Keywords: [F-18] FDDNP-PET; Alzheimer's disease (AD); beta amyloid; tau; positron emission tomography; chronic traumatic encephalopathy (CTE); traumatic encephalopathy syndrome (TES)
MeSH Terms: conditions — Alzheimer Disease; Plaque, Amyloid; Pick Disease of the Brain; Chronic Traumatic Encephalopathy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood tests will be performed for safety assessment. Tests performed include:
  * Complete Blood Count with Differential
  * Free T4 Index
  * Vitamin B12 Serum
  * Chemistry Panel
  * Uric Acid
  * Thyroid-Stimulating Hormone
  * Cholesterol
  * Genetic Testing (APoE status)
  For participants that consent to autopsy, the following procedures will be performed:
  • At the time of death, the brain will be harvested within a 24 hour postmortem interval by standard autopsy procedures. The brain will be preserved, rinsed and dissected for the collection of regions of interest (ROIs) adapted and modified from the National Institute on Aging (NIA)- Alzheimer's Association guidelines for the neuropathologic assessment of AD (Hyman et al, 2012).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Suspected AD: Participants with suspected AD enrolling in the trial must meet all of the following criteria:
  * Cognitive deficits do not occur exclusively in the context of a delirium.
  * Cognitive deficits are not better explained by another mental disorder (e.g., major depressive disorder, schizophrenia).
  * There is insidious onset and gradual progression of impairment in one or more cognitive domains.
  * The participant has documented memory problems in one or more other cognitive domains, such as language, visual-spatial functioning, executive functioning, etc. (Busse et al., 2006).
  Interventions: Biological: [F-18]FDDNP-PET
- Suspected CTE / TES: Required Features:
  * Persistence of symptoms for longer than 2 years; no other neurologic disorder that is more likely to account for all the clinical features; history of head trauma exposure; progressive course; and at least 1 supportive feature
  * History of head trauma exposure, typically associated with history of concussion, although may be limited to subconcussive trauma
  * Head trauma exposure is repetitive in nature
  * Demonstrated progressive course
  * Delayed symptom onset
  * Self-report or observer report of cognitive dysfunction, confirmed with objective cognitive decline documented by results of formal neuropsychological testing. Cognitive decline typically affects more than 1 domain (executive, visuospatial, memory, and language).
  Supportive Features (only 1 required):
  * Emotional dysregulation
  * Behavioral change
  * Motor disturbance
  Interventions: Biological: [F-18]FDDNP-PET

INTERVENTIONS:
Biological: [F-18]FDDNP-PET — [F-18]FDDNP, or 2-(1-{6-[(2-[F-18]fluoroethyl)(methyl)amino]-2- naphthyl}ethylidene)malononitrile, is a positron emission tomography (PET) radiotracer developed for the in vivo visualization of tau and amyloid-beta (Aβ) deposition in the brain.

SUMMARY:
The primary objective of this study is to demonstrate the safety and efficacy of positron emission tomography (PET) imaging with a radioactive compound called [F-18]FDDNP in subjects with suspected Alzheimer's disease or suspected chronic traumatic encephalopathy (CTE) to predict clinical decline after one and two years.

DETAILED DESCRIPTION:
The investigators will enroll approximately 180 participants with mild cognitive impairment (90 with suspected Alzheimer's Disease and 90 with suspected Chronic Traumatic Encephalopathy with a history of head trauma).

Participants will come to UCLA for 4 visits and will be called twice. The study duration is 2 years.

Participants will first complete an over the phone screening to assess their eligibility. If they pass the phone screen, then they will be invited to complete an in-person screen and will sign the informed consent form. They will then undergo a neurological evaluation, blood draw, and neuropsychological testing.

Within a month of the screening visit, participants will complete the imaging visit. Participants will undergo a magnetic resonance imaging (MRI) scan, if eligible, and a PET scan with FDDNP. For participants who are unable to undergo an MRI due to contraindications, they will complete a CT scan.

Participants will be monitored for possible adverse events following the procedures and will be called 24 hours later and 2 weeks later to assess for any potential adverse events.

At the one and two-year follow-up visits, participants' medical history will be reviewed. At this time, they will also complete a neuropsychiatric evaluation, blood draw and neuropsychological testing.

Prediction of clinical and cognitive decline from [F-18] FDDNP PET scan readers (blinded to clinical evaluations) and clinicians (blinded to [F-18]FDDNP PET scan results) will be compared with actual clinical outcomes determined at one and two-year follow-up visits.

ELIGIBILITY:
Inclusion criteria for all participants

Participants enrolling in the trial must meet all of the following criteria:

* Participant may be male or female and of any race/ethnicity
* Age 18 to 80 years at the time of study drug dosing
* Female participants must be either surgically sterilized or post-menopausal, defined as at least one-year without menses as reported by the participant or have a negative serum pregnancy test
* Participant or participant's legally acceptable representative (when appropriate) provides informed consent
* Participant is capable of complying with study procedures
* Participant is capable of communicating with study personnel
* Participant is willing to undergo longitudinal follow-up at 1 and 2 years after the Imaging Visit
* All participants will meet criteria for mild cognitive impairment (Petersen et al, 2014) or Mild Neurocognitive Disorder (APA, 2013):
* Patient awareness of a memory problem, preferably confirmed by another person who knows the patient
* Memory impairment detected with standard assessment tests
* Ability to perform normal daily activities
* For a broad definition of mild cognitive impairment, we also use guidelines to identify those with other mild cognitive impairment subtypes, including those with memory impairment and/or additional cognitive deficits (Winblad et al, 2004). The diagnosis will be corroborated by clinical judgment and include participants who score 1 standard deviation or more below the age-corrected norms because this threshold for impairment yields high sensitivity for predicting dementia (de Jager et al, 2005). To balance increased sensitivity with specificity, impairment on at least 2 neuropsychological tests will be required (Jak et al., 2009).

Inclusion criteria for participants with suspected CTE

Participants with suspected CTE enrolling in the trial must meet all of the following criteria:

• Participant must meet the most recently proposed clinical criteria for suspected CTE (termed possible traumatic encephalopathy syndrome or TES; Reams et al, 2016). These proposed diagnostic criteria for possible TES include the following features:

Required Features:

* Persistence of symptoms for longer than 2 years; no other neurologic disorder that is more likely to account for all the clinical features; history of head trauma exposure; progressive course; and at least 1 supportive feature
* History of head trauma exposure, typically associated with history of concussion, although may be limited to subconcussive trauma
* Head trauma exposure is repetitive in nature
* Demonstrated progressive course
* Delayed symptom onset
* Self-report or observer report of cognitive dysfunction, confirmed with objective cognitive decline documented by results of formal neuropsychological testing. Cognitive decline typically affects more than 1 domain (executive, visuospatial, memory, and language).
* Supportive Features (only 1 required):
* Emotional dysregulation: including depression, anxiety, agitation, aggression, paranoid ideation, deterioration of interpersonal relationships, and suicidality
* Behavioral change: including violence, poor impulse control, socially inappropriate behavior, avolition, apathy, change in personality, and comorbid substance abuse
* Motor disturbance: including bradykinesia, tremor, rigidity, gait instability, dysarthria, dysphagia, and ataxia

Inclusion criteria for participants with suspected AD

Participants with suspected AD enrolling in the trial must meet all of the following criteria:

* Cognitive deficits do not occur exclusively in the context of a delirium.
* Cognitive deficits are not better explained by another mental disorder (e.g., major depressive disorder, schizophrenia).
* There is insidious onset and gradual progression of impairment in one or more cognitive domains.
* The participant has documented memory problems in one or more other cognitive domains, such as language, visual-spatial functioning, executive functioning, etc. (Busse et al., 2006).

Exclusion criteria for all participants

Participants meeting any of the following criteria will not be enrolled in the study:

* Participant is pregnant or nursing
* Phone screen of Telephone Interview for Cognitive Status-modified (TICS-M) ≥ 33
* Participant unable to remain still for duration of imaging procedure or has an inability to tolerate neuropsychological, clinical, or PET scan studies (e.g., head tremor that may cause head motion artifact, uncontrollable psychosis, acute suicidality)
* Participant has prior history of stroke or other condition of the head or neck that, in the investigator's opinion, might affect circulation to the head or image interpretation
* Preexisting major neurologic or other physical illness that could confound results (e.g., multiple sclerosis, diabetes, cancer)
* Participant has a major psychiatric disorder such as mania or schizophrenia, which might interfere with completing study procedures (APA, 2013)
* Participant has a psychiatric disorder, such as anxiety or depression, severe enough to interfere with completing study procedures
* Participant has a condition or personal circumstance that, in the judgment of the investigator, might interfere with the collection of complete accurate quality data
* Participant has a history of significant prescription drug, non-prescription drug, or alcohol abuse, including but not limited to marijuana, cocaine, heroin or derivatives
* Participant has previously received [F-18]FDDNP at any time, or any other investigational product within the past thirty days
* Participant has a history of allergic reactions to albumin
* Participant has severe anemia in which case the use of albumin would be medically contraindicated
* Participant has cardiac failure in which case the use of albumin would be contraindicated
* Participant has unstable cardiac disease or uncontrolled hypertension (systolic BP > 170 or diastolic BP > 100)
* Participants taking ibuprofen or naproxen will be asked to stop taking the medication for five days before the PET scan since these medicines may affect [F-18]FDDNP-PET scan results. Other anti-inflammatory medicines, such as diclofenac or aspirin, can be substituted during that period. If the participant cannot temporarily discontinue the medicine, that participant will be excluded from the study
* Participant has used of any investigational drugs within the previous month or has participated in imaging or other clinical research protocols that might confound study results

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will recruit participants with mild cognitive impairment and suspected CTE or suspected AD.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-05 (Estimated); Primary Completion 2021-05-03 (Actual); Study Completion 2021-05-03 (Actual)

PRIMARY OUTCOMES:
Clinical Dementia Rating Sum of Box Scores (CDR-SB) | 2 years
  We propose to use the CDR Sum of Box Scores (CDR-SB) as the primary efficacy endpoint to be predicted (at two-year follow-up) following baseline when the [F-18]FDDNP-PET imaging is performed. The CDR-SB score is obtained by summing each of the domain box scores, with scores ranging from 0 to 18. We will use change in CDR-SB score as the common outcome variable. We will convert individual CDR-SB scores into standardized scores by subtracting the baseline mean and dividing by the baseline standard deviation of the study sample (Monsell et al, 2012). Individuals experiencing worsening of cognition by at least 0.5 standard deviation per year in the standardized CDR-SB score will be classified as cognitive decliners; others will be classified as cognitive maintainers.

SECONDARY OUTCOMES:
Change in Executive Functioning Domain Score | 2 years
  Calculated as the average of z- transformed scores of: Trails B-A, Category Fluency, Letter Fluency, and Wechsler Adult Intelligence Scale-IV Digit Symbol and Digit Span backwards (Harrison et al., 2007).
Conversion to Dementia | 2 years
  For a dementia diagnosis, we will use major neurocognitive disorder according to the Diagnostic and Statistical Manual-5 [DSM-5] criteria (APA, 2013; Csukly et al, 2016).

CONTACTS AND LOCATIONS:
Overall Officials: Helen Lavretsky, MD, Principal Investigator — University of California, Los Angeles, Semel Institute

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: ICF, CSR

REFERENCES:
- [Background] American Psychiatric Association. Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5). Washington, DC: American Psychiatric Association, 2013.
- [Background] Busse A, Hensel A, Guhne U, Angermeyer MC, Riedel-Heller SG. Mild cognitive impairment: long-term course of four clinical subtypes. Neurology. 2006 Dec 26;67(12):2176-85. doi: 10.1212/01.wnl.0000249117.23318.e1. PMID 17190940
- [Background] Csukly G, Siraly E, Fodor Z, Horvath A, Salacz P, Hidasi Z, Csibri E, Rudas G, Szabo A. The Differentiation of Amnestic Type MCI from the Non-Amnestic Types by Structural MRI. Front Aging Neurosci. 2016 Mar 30;8:52. doi: 10.3389/fnagi.2016.00052. eCollection 2016. PMID 27065855
- [Background] de Jager CA, Budge MM. Stability and predictability of the classification of mild cognitive impairment as assessed by episodic memory test performance over time. Neurocase. 2005 Feb;11(1):72-9. doi: 10.1080/13554790490896820. PMID 15804927
- [Background] Harrison J, Minassian SL, Jenkins L, Black RS, Koller M, Grundman M. A neuropsychological test battery for use in Alzheimer disease clinical trials. Arch Neurol. 2007 Sep;64(9):1323-9. doi: 10.1001/archneur.64.9.1323. PMID 17846273
- [Background] Hyman BT, Phelps CH, Beach TG, Bigio EH, Cairns NJ, Carrillo MC, Dickson DW, Duyckaerts C, Frosch MP, Masliah E, Mirra SS, Nelson PT, Schneider JA, Thal DR, Thies B, Trojanowski JQ, Vinters HV, Montine TJ. National Institute on Aging-Alzheimer's Association guidelines for the neuropathologic assessment of Alzheimer's disease. Alzheimers Dement. 2012 Jan;8(1):1-13. doi: 10.1016/j.jalz.2011.10.007. PMID 22265587
- [Background] Jak AJ, Bondi MW, Delano-Wood L, Wierenga C, Corey-Bloom J, Salmon DP, Delis DC. Quantification of five neuropsychological approaches to defining mild cognitive impairment. Am J Geriatr Psychiatry. 2009 May;17(5):368-75. doi: 10.1097/JGP.0b013e31819431d5. PMID 19390294
- [Background] Monsell SE, Liu D, Weintraub S, Kukull WA. Comparing measures of decline to dementia in amnestic MCI subjects in the National Alzheimer's Coordinating Center (NACC) Uniform Data Set. Int Psychogeriatr. 2012 Oct;24(10):1553-60. doi: 10.1017/S1041610212000452. Epub 2012 Apr 16. PMID 22717299
- [Background] Petersen RC, Caracciolo B, Brayne C, Gauthier S, Jelic V, Fratiglioni L. Mild cognitive impairment: a concept in evolution. J Intern Med. 2014 Mar;275(3):214-28. doi: 10.1111/joim.12190. PMID 24605806
- [Background] Reams N, Eckner JT, Almeida AA, Aagesen AL, Giordani B, Paulson H, Lorincz MT, Kutcher JS. A Clinical Approach to the Diagnosis of Traumatic Encephalopathy Syndrome: A Review. JAMA Neurol. 2016 Jun 1;73(6):743-9. doi: 10.1001/jamaneurol.2015.5015. PMID 27111824
- [Background] Winblad B, Palmer K, Kivipelto M, Jelic V, Fratiglioni L, Wahlund LO, Nordberg A, Backman L, Albert M, Almkvist O, Arai H, Basun H, Blennow K, de Leon M, DeCarli C, Erkinjuntti T, Giacobini E, Graff C, Hardy J, Jack C, Jorm A, Ritchie K, van Duijn C, Visser P, Petersen RC. Mild cognitive impairment--beyond controversies, towards a consensus: report of the International Working Group on Mild Cognitive Impairment. J Intern Med. 2004 Sep;256(3):240-6. doi: 10.1111/j.1365-2796.2004.01380.x. PMID 15324367